CLINICAL TRIAL: NCT05586867
Title: Study of Markers of Iron Metabolism and Their Relationship With Phosphocalcic and Hepatic Metabolism and Inflammation in Hemodialysis Patients
Acronym: MARMEFE
Status: Recruiting | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01329-32
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Iron Metabolism Disorders; Calcium Phosphate Metabolism; Hepatic Metabolic Disorders; Hemodialysis Complication
MeSH Terms: conditions — Iron Metabolism Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodialysis patient
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — 15 mL of blood to follow the evolution of hepcidin and erythroferrone levels

SUMMARY:
From a scientific point of view and for publication purposes, it therefore seems important to study the metabolism of iron and in particular to define its conditions of absorption, metabolism, elimination and storage in the body at course of advanced renal failure.

The study will follow the evolution of hormones regulating iron metabolism and put into perspective their links with phosphocalcic and hepatic metabolisms as well as inflammation in hemodialysis patients.

The main objective of this program is to study the evolution of hepcidin and erythroferrone levels in hemodialysis patients. These two biomarkers regulating iron metabolism are not performed routinely in dialysis centers and are not listed in the nomenclature.

ELIGIBILITY:
Inclusion Criteria:

* Adult dialysis patient
* Patient able to understand the information necessary for the study and having signed his written consent to participate
* Affiliated patient or beneficiary of a social security scheme.

Exclusion Criteria:

* Medically unstable or frail patient
* Patient with hemoglobin less than 7g/dl
* Patient with HIV+ or AIDS, patient with replicating hepatitis B or C
* Patient participating in another clinical study requiring an additional blood sample
* Patient benefiting from legal protection measures (guardianship, guardianship, etc.) adult under guardianship, guardianship or other legal protection, deprived of freedom by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis adult patient
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
concentration of the two main markers concerning iron metabolism: hepcidin (ng/ml) and erythroferone (ng/ml). | 5 years
  These will be dosed twice over a year of dialysis and for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France